CLINICAL TRIAL: NCT04175158
Title: A Randomized, Double-blind, Parallel-controlled Comparative Study to Evaluate the PK Pharmacokinetic Similarity After Single Administration of GB222 and Bevacizumab in Healthy Volunteers.
Brief Title: Clinical Trial in Chinese Healthy Volunteers of GB222
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENOR GB222-001; V1.3
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB222 (Experimental): 1mg/kg
  Interventions: Biological: GB222
- Bevacizumab (Active Comparator): 1mg/kg
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: GB222 — Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection Injection; strength 100mg/4ml/bottle; intravenous drip; a total of one administration, dosage 1mg/kg; The 2.5ml syringe is used to collect required volume of the drug, and then it will be added to 250 ml of 0.9% sodium chloride solution. The infusion bag should be gently inverted to prevent air bubbles. If the required volume is > 2.5 ml, it should be collected twice, 2.5ml for the first time and the rest for the second time.
  Other Names: Recombinant humanized antivascular endothelial growth factor monoclonal antibody injection
  Arms: GB222
Biological: Bevacizumab — Injection; strength 100mg/4ml/bottle; intravenous drip; a total of one administration, dosage 1mg/kg; The 2.5ml syringe is used to collect required volume of the drug, and then it will be added to 250 ml of 0.9% sodium chloride solution. The infusion bag should be gently inverted to prevent air bubbles. If the required volume is > 2.5 ml, it should be collected twice, 2.5ml for the first time and the rest for the second time.
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
The primary objective of this study is to evaluate the similarity of the primary pharmacokinetic (PK) parameter AUC0-t of GB222 and bevacizumab after single administration; the secondary objective is to observe the safety and similarities and safety of other pharmacokinetic (PK) parameters (Cmax, AUC0-∞ etc.) and immunogenicity of GB222 and bevacizumab after single administration.

ELIGIBILITY:
1. Subjects who voluntarily participated in the clinical study and sign the informed consent form;
2. Healthy male adult volunteers aged 18 to 45 years;
3. The subjects have qualified physical examination within 28 30 days before the study, the body mass index (BMI) is within the range of 19.0~24.0, 50kg for males³ and 45kg for females³, the body weight of males and females is not more than 75kg (inclusive);
4. The subjects agree and adopt reliable contraceptive methods to ensure that they have no pregnancy plain from the beginning of the study to 6 months after the end of this study;
5. Based on physical examination, medical history, vital signs, electrocardiogram, etc., the researchers determined that the body condition of participant was good;
6. The subjects can well communicate with the investigators and complete the study as required by the study.

Exclusions：

1. Allergic constitution; known allergic to the components of the investigational product or allergy history to any drug or food or pollen; subjects who have abnormal serum immunoglobulin E (IgE);
2. Any current signs and symptoms or abnormalities in laboratory tests may indicate acute or subacute infection (fever, cough, urination, pain, abdominal pain, diarrhea, skin infection, wound, etc.)
3. History of drug addiction or drug abuse; subjects with positive urine drug screening;
4. Clear medical history of central nervous system, cardiovascular, renal, hepatic, gastrointestinal, respiratory, metabolic system or other significant diseases; medical history of hypertension or screening systolic blood pressure³ of 140mmHg and/or diastolic blood pressure³ of 90mmHg,which are clinically significant at the discretion of the investigators;
5. People with malignant tumors;
6. Participated in other clinical studies within 3 months before enrollment, or subjects who received drugs which are known to injure the major organs within 3 months before enrollment;
7. Blood donation within 3 months before enrollment;
8. Surgery operation within 3 months before enrollment;
9. Use of prescription drugs or non-prescription drugs within 14 days before enrollment;
10. ALT or AST>1.5 ULN, Cr>ULN;
11. Hematology test: WBC<3.0×10 9 /L or > 9.5×10 9 /L; ANC < 1.5×10 9 /L; PLT<100×10 9/L; HGB<104 g/L,conform to any of these items;
12. Any of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
13. Subjects who have positive anti-drug antibody (ADA);
14. Positive tumor marker (CEA、AFP、PSA、CA-125);
15. Abnormal coagulation function, which is judged by the researcher to be clinically significant;
16. Patients with a previous history of digestive tract ulcer, cerebrovascular accident, vascular lesions, etc., currently have open wounds of skin and mucosa. The researchers considered that other volunteers with risk of bleeding or coagulation should not be included in the study
17. Patients with a history of mental illness.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male only
Enrollment: 84 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
AUC 0- t | Up to 84 days
  AUC 0- t

SECONDARY OUTCOMES:
Cmax | Up to 84 days
  Cmax
AUC0-∞ | Up to 84 days
  AUC0-∞
ADA | Up to 84 days
  ADA

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, Master, Principal Investigator — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No